CLINICAL TRIAL: NCT03526809
Title: A Physiological Study of the Metabolism of Pyruvate in High Grade Serous Ovarian Cancer Using Hyperpolarised Carbon-13 Magnetic Resonance Spectroscopic Imaging
Brief Title: Molecular Imaging and Spectroscopy With Stable Isotopes in Oncology and Neurology
Acronym: MISSION-ovary
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Surrin Deen, Honorary Clinical Fellow, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: A093768
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Ovarian Cancer
Keywords: Magnetic resonance imaging
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fixed and frozen ovarian cancer specimens from areas imaged collected by image guided biopsy and surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ovarian cancer patients: MRI and FDG-PET imaging
  Interventions: Diagnostic Test: MRI scan and FDG-PET scan

INTERVENTIONS:
Diagnostic Test: MRI scan and FDG-PET scan — Scanning with MRI and FDG-PET

SUMMARY:
Patients with known ovarian cancer will be imaged up to four times with FDG-PET, C13 MRI and other novel MRI techniques during their treatment course including: before the start of any treatment (with optional repeat scanning), after the first dose of chemotherapy (optional), after the third dose of chemotherapy (optional) and after surgery (optional). Imaging findings will be compared to biological properties of cancer tissue samples.

DETAILED DESCRIPTION:
This is a single-centre prospective physiological study.

1. Participants will be recruited through MDTs and clinics.
2. Baseline screening blood tests will be performed.
3. Baseline MRI will be undertaken to identify lesions to be studied. This will be followed by hyperpolarised carbon-13 MRSI after the injection of hyperpolarised 13C-pyruvate. Scanning with 18F-FDG PET in combination with CT or MRI may optionally be performed in the same imaging visit.
4. A subset of patients (up to 10) will undergo repeat hyperpolarised carbon-13 MRSI within 5 days of baseline imaging to assess for reproducibility of the imaging test.
5. Where possible, image-guided biopsy will be performed to obtain tissue from selected lesions for analysis.
6. During the first month of and later during systemic anticancer therapy, MRI and carbon-13 MRSI will be again carried out to assess to look for changes in pyruvate metabolism. If possible, a further biopsy will be undertaken at this stage. Scanning with 18F-FDG PET in combination with CT or MRI may optionally be performed in the same imaging visit.
7. MRI and carbon-13 MRSI will be carried out after the full course of systemic anticancer therapy, to assess for treatment response and to identify lesions in preparation for tissue extraction at surgery. Scanning with 18F-FDG PET in combination with CT or MRI may optionally be performed in the same imaging visit.
8. During surgery, tissue samples will be collected either by excision or biopsy.
9. MRI may be performed after surgery in selected patients.
10. In up to 10 participants, carbon-13 MRSI will be done 3 to 6 weeks after surgery to look for areas of pyruvate or lactate accumulation that may correlate with long term prognosis. Only participants who are not part of the subset undergoing retest carbon-13 MRSI to assess for reproducibility will be invited for post-surgical carbon-13 MRSI, this is to keep the number of carbon-13 MRSI scans each participant has at a maximum of four in order to minimise inconvenience to participants caused by having to make repeat visits for imaging.
11. Participants will be followed up for one year in the clinic and/or through their GP.

ELIGIBILITY:
Inclusion Criteria:

* To be included in this study the patient must:

  1. Be 18 years or older.
  2. Have a confirmed or likely diagnosis of HGSOC, breast cancer, prostate cancer, pancreatic mass, liver mass, renal mass or brain tumour.
  3. Be aware of their diagnosis.
  4. Be a likely surgical candidate who is fit for possible surgery.
  5. Have no contraindications to the use of the IV contrast agents involved in this study.
  6. Be able to provide written informed consent according to ICH/GCP, national and local regulations.
  7. Volunteers of childbearing potential must have a negative pregnancy test, either urinary or blood prior to enrolment.
  8. Have ECOG performance status 0 or 1.
  9. Express willingness and ability to comply with scheduled visits, laboratory tests, imaging and other study procedures.

Exclusion Criteria:

* The presence of any of the following will preclude the patient from the study:

  1. Any disorder that may adversely affect levels of pyruvate or lactate such as diabetes mellitus.
  2. The use of medications that may affect levels of pyruvate or lactate such as metformin or insulin.
  3. Known allergy or adverse reaction to any of the injected contrast agents proposed for use in this study.
  4. Pregnancy or breastfeeding.
  5. Other severe acute or chronic medical or psychiatric conditions that may increase the risk associated with study participation or in the judgement of the investigators make it undesirable for the patient to enter the study.
  6. Laboratory abnormalities that may have an unknown or unpredictable impact on study results.
  7. Not suitable for MR scanning e.g. severe obesity, inability to lie still or contraindicated metal implants such as the intrauterine contraceptive device.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patient with ovarian cancer
Study Population: Patients with ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Imaging of the metabolism of hyperpolarized 13C-pyruvate in ovarian cancer tissue to hyperpolarized 13C-lactate. | 1 July 2016 to 31 December 2018
  Imaging of the metabolism of hyperpolarized 13C-pyruvate in ovarian cancer tissue to hyperpolarized 13C-lactate.

SECONDARY OUTCOMES:
Correlation of the hyperpolarized 13C images from tumour with histological, biochemical and genetic information gained after surgery and/or biopsy. | 1 July 2016 to 31 December 2018
  Correlation of the hyperpolarized 13C images from tumour with histological, biochemical and genetic information gained after surgery and/or biopsy.
Detection of the change in the metabolism of hyperpolarized 13C-pyruvate following systemic anticancer therapy. | 1 July 2016 to 31 December 2018
  Detection of the change in the metabolism of hyperpolarized 13C-pyruvate following systemic anticancer therapy.

OTHER OUTCOMES:
To determine if the metabolism of hyperpolarized 13C-pyruvate can be detected in a small number of patients with breast cancer, prostate cancer, pancreatic masses, liver masses, renal masses and brain tumours | 1 July 2016 to 31 December 2018
  To determine if the metabolism of hyperpolarized 13C-pyruvate can be detected in a small number of patients with breast cancer, prostate cancer, pancreatic masses, liver masses, renal masses and brain tumours
To investigate the relationship between hyperpolarized 13C-pyruvate MRSI and 18F-FDG uptake on PET. | 1 July 2016 to 31 December 2018
  To investigate the relationship between hyperpolarized 13C-pyruvate MRSI and 18F-FDG uptake on PET.

CONTACTS AND LOCATIONS:
Locations (1):
- Addenbrooke's Hospital, Cambridge, Please Select An Option Below, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Consent has been obtained to share imaging results with other researchers working in similar imaging however there are no definite plans to do this unless results require verification from other sites.